CLINICAL TRIAL: NCT06909851
Title: Comparison of the Effectiveness of Adductor Canal Block and Genicular Nerve Block on Postoperative Pain and Analgesic Use in Arthroscopic Knee Surgeries
Brief Title: Comparison of Pain Relief After Arthroscopic Knee Surgery: Adductor Canal Block and Genicular Nerve Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, Associate Professor Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSH-ANES-SA-01
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use; Pain Postoperative; Arthroscopic Knee Surgeries
Keywords: Genicular Nerve Block; Arthroscopic Knee Surgery; Adductor Canal Block; Postoperative Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients who are admitted to the orthopedic and traumatology clinic and are scheduled for arthroscopic knee surgery will be informed and monitored prior to the operation under spinal anesthesia. Preoperatively, either Adductor Canal Block (ACB) (Group A) or Genicular Nerve Block (GNB) (Group B) will be applied. Randomization will be performed using a computer-based method (http://www.randomizer.org) with a 1:1 allocation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACB Group (Active Comparator): Participants undergoing arthroscopic knee surgery under spinal anestesia receiving pre operative Adductor Canal Block (ACB)
  Interventions: Procedure: Adductor Canal Block (ACB)
- Genicular Nerve Block (Active Comparator): Participants undergoing arthroscopic knee surgery under spinal anestesia receiving pre operative Genicular Nerve Block (GNB)
  Interventions: Procedure: Genicular Nerve Block (GNB)

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) — Evaluation of postoperative analgesic effectiveness of ACB block in participants undergoing arthroscopic knee surgery under spinal anesthesia.
  Arms: ACB Group
Procedure: Genicular Nerve Block (GNB) — Evaluation of postoperative analgesic effectiveness of GNB block in participants undergoing arthroscopic knee surgery under spinal anesthesia.
  Arms: Genicular Nerve Block

SUMMARY:
This prospective randomized study aims to compare the analgesic efficacy of Adductor Canal Block (ACB) and Genicular Nerve Block (GNB) groups to relieve postoperative pain in participants between ages of 18-72 undergoing arthroscopic knee surgery under spinal anesthesia. The main question it aims to answer is:

To demonstrate whether Adductor Canal Block or Genicular Nerve Block is more effective in postoperative analgesia in patients undergoing arthroscopic knee surgery based on pain scores, opioid consumption and patient satisfaction.

Arthroscopic knee surgeries cause severe pain especially with movement in the post-operative period. After surgery, the movements of the participants are severely restricted because of pain, which increases the possibility of complications and postpones post-operative knee exercises. In this study, the participants' pain status, VAS score, opioid consumption and patient satisfaction will be measured with a simple scoring system for 24 hours at predetermined time points and then compared. Both types of blocks have pain-relieving effects. This study will only investigate which one is more effective in reducing pain, and there will be no deficiency in relieving the pain of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary willingness to participate in the study.
* Patients undergoing arthroscopic knee surgery (meniscus, ACL, arthroscopic intervention etc).
* ASA I-II-III classification.
* Aged between 18-72 years.
* No contraindications for regional anesthesia, and deemed suitable for regional anesthesia by the anesthesiologist.
* Undergoing surgery under spinal anesthesia.
* Fully oriented and able to cooperate.

Exclusion Criteria:

* Undergoing surgery under general anesthesia.
* Chronic analgesic use.
* Presence of an active infection at the procedure site.
* Outside the appropriate age range.
* Inability to comply with postoperative pain/NRS follow-ups.
* ASA IV-V classification.
* Non-voluntary patients.
* Pregnancy.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness on Pain Scores (NRS) | Postoperative 24 hours
  Postoperative pain assessment is performed using the Numerical Rating Scale (NRS). Participants are asked about their rest pain at Baseline 0, postoperative 1st, 2nd, 4th, 6th, 12th, and 24th hours after applying a preoperative peripheral nerve block. With this method, participants rate their pain with a precise numerical value from 0 to 10. While zero(0) represents "no pain"; Ten (10) represents the opposite end of the pain continuum (e.g., "The most intense pain imaginable," "As intense pain as possible," "Maximum pain").

SECONDARY OUTCOMES:
Amount of rescue analgesia administration | Postoperative 24 hours.
  After the surgery all patients will be given 4 times a day Paracetamol 1 gram. Patients who still have pain (NRS 4 or higher) will be given Tramadol 1 mg/kg (maximum 400 mg Tramadol daily). Postoperative 24 hours the amount of the rescue analgesic (Tramadol) will be noted.
Postoperative Blood pressure | Postoperative 24 hours
  Participants' blood pressure (mm/hg) will be monitored for 24 hours (Post op 1st, 2nd, 4th, 6th, 12th and 24th hours) postoperatively.
Length of hospital stay | Postoperative 14 days
  Length of hospital stay will be noted.
First Time Of Mobilisation/Exercise | Postoperative 24 hours
  First time of mobilisation/exercise will be noted.
The Time of Rescue Analgesic | Postoperative 24 hours
  After the surgery all patients will be given 4 times a day Paracetamol 1 gram. Patients who still have pain (NRS 4 or higher) will be given Tramadol 1 mg/kg (maximum 400 mg Tramadol daily). Postoperative 24 hours the time of the rescue analgesic usage (Tramadol) will be noted.
Postoperative heart rate | Postoperative 24 hours
  Participants' heart rate (bpm) will be monitored for 24 hours (Post op 1st, 2nd, 4th, 6th, 12th and 24th hours) postoperatively.
Postoperative oxygen saturation levels | Postoperative 24 hours
  Participants' oxygen saturation levels (spO2 %) will be monitored for 24 hours (Post op 1st, 2nd, 4th, 6th, 12th and 24th hours) postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam & Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vora MU, Nicholas TA, Kassel CA, Grant SA. Adductor canal block for knee surgical procedures: review article. J Clin Anesth. 2016 Dec;35:295-303. doi: 10.1016/j.jclinane.2016.08.021. Epub 2016 Oct 11. PMID 27871547
- [Background] Tamam A, Guven Kose S, Kose HC, Akkaya OT. Comparison of the Effectiveness of Ultrasound-Guided Proximal, Mid, or Distal Adductor Canal Block after Knee Arthroscopy. Turk J Anaesthesiol Reanim. 2023 Apr;51(2):135-142. doi: 10.5152/TJAR.2023.22225. PMID 37140579